CLINICAL TRIAL: NCT00861172
Title: Longitudinal (Weekly) Follow-up of Active Plaques in Multiple Sclerosis With 3 Teslas Multi-modality MRI Using Diffusion, Perfusion, Venography and Proton Spectroscopy
Acronym: IRM 3T-SEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Pr. Francois COTTON, Hospices Civils de Lyon
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2008.532
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Lesions; Multiple Sclerosis
Keywords: Multiple sclerosis; Active plaque; Multimodal analysis; 3T MRI; Weekly follow-up; Physiopathology; Physiopathology of active lesions formation in Multiple Sclerosis using multimodal MR sequences
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: 3T MR scanner

INTERVENTIONS:
Procedure: 3T MR scanner — The follow-up will be scheduled for one year; it will consist in a weekly MR examination during the first two months, and subsequently on the 6th and the 12th months.
  We will perform for each MRI exploration an intravenous injection of contrast agents: gadobutrol (gadovist 1,0 mmol/ml) which is a stable agent with a cyclic structure. This agent is few responsible for NFS, given their low capacity to liberate gadolinium GD3+ in tissues.
  The same imaging protocol will be performed for each MR examination. Evaluation of creatinemia will be used before inclusion and during the 1st, 3rd, 5th, 7th, 9th, and the 10th MRI examination. Thus we will take advantage of catheter to perform the creatinemia blood test and to reduce the discomfort produced by the injection.

SUMMARY:
It is difficult to determinate prognostic criteria of Multiple Sclerosis with conventional MRI insofar as physiopathology is not well-known: the precise sequences of events leading to plaque formation and axonal injury are still not completely understood.

Some elements involved in plaque formation can be studied thanks to MR techniques (cerebrospinal fluid and periveinular spaces, neuronal injury, microglia, and cerebral microcirculation's dysfunction).

This study aims at giving a better understanding of MS plaques' physiopathology, using data from modern MRI through a longitudinal followed up with weakly MR 3T examination.

DETAILED DESCRIPTION:
The objective of this work are:

* study weakly development of the active MS plaque with multimodal MRI parameters using advanced MRI techniques: Veinography/3D FLAIR, Diffusion (CDA), Perfusion (CBV, CBF, MTT) MR Spectroscopy (NAA, myo-inositol, choline, lactate…) and enhanced 3DT1 sequences.
* define prognostic markers of MS aggressiveness ("black holes")
* Study development of MS plaque around venous structures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Health coverage.
* Any form of MS defined by Mc Donald's criteria (2005).
* Patients having shown an enhanced plaque on a less than six month MRI examination.

Exclusion Criteria:

* Patients with an immunomodulating therapy like natalizumab (Tysabri) and intravenous immunosuppressive therapies. Other therapies will not be excluded from this study. For patients treated by systemic corticotherapy, a one-month delay will be necessary before a MRI examination.
* Cerebral microangiopathy (diabetes, arterial hypertension, vascularitis…)
* Patient with classical MRI contraindication like pace-maker, cardiac valvulosis, claustrophobia, allergy to contrast agent …
* Pregnancy or pregnancy desire.
* Patient with a low creatinine clearance <60 ml/mn

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Modification of MR parameters before and after the blood brain barrier disruption observed in newly enhancing lesion in MS. | each week for 2 months, at 6 month and at 12 month

SECONDARY OUTCOMES:
Predictive scorers of plaque transformation in "black-holes", which correspond with a pejorative evolution of accurate lesions, also defined by a focal destruction of cerebral tissue. | each week for 2 months, at 6 month and at 12 month
Relation between plaques development and cerebral venous structures. | each week for 2 months, at 6 month and at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Francois Cotton, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Services de Neurologie A et Service de Neuroradiologie, Pôle transversal d'imagerie, Hôpital Neurologique, Bron, France

REFERENCES:
- [Derived] Hannoun S, Roch JA, Durand-Dubief F, Vukusic S, Sappey-Marinier D, Guttmann CR, Cotton F. Weekly multimodal MRI follow-up of two multiple sclerosis active lesions presenting a transient decrease in ADC. Brain Behav. 2015 Feb;5(2):e00307. doi: 10.1002/brb3.307. Epub 2015 Jan 16. PMID 25642392